CLINICAL TRIAL: NCT01395576
Title: Evaluation of the Genu Neurexa Orthosis in Post Stroke Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: statistical significance of the results was reached for the 34 subjects who participated in teh study.
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Otto Bock Healthcare Products GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GENU-HMO-CTIL
Record Dates: First submitted 2011-07-03; First posted 2011-07-15 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2012-10

CONDITIONS: Stroke
Keywords: Genu recurvatum; Knee hyper extension; Orthosis; Gait analysis; Post stroke
MeSH Terms: conditions — Stroke

INTERVENTIONS:
Device: Genu Neurexa orthosis — Knee orthosis for the prevention of knee hyper extension

SUMMARY:
Post stroke patients often suffer from decrease in strength, loss of balance and gait asymmetry. Accordingly, these patients are at high risk for falls and fall-related injury. The presence of spastic or retracted muscles, e.g. the ankle plantar flexors or the quadriceps in combination with hamstrings weakness, causes knee hyperextension, which increases the stance phase duration and makes it difficult to achieve symmetrical gait. Additionally, this gait disorder can be painful as a result of stress to the ligaments and tendons at the posterior aspect of the knee.

The Genu Neurexa orthosis is designed to stabilize the knee, enable balance control and prevent hyperextension. In order to assess the effect of the orthosis on the gait and balance characteristics of stroke patients the investigators will conduct subjective patient's satisfactory questionnaire, complete physical and functional evaluation and gait analysis, as well as dynamic electromyography (EMG) muscle activation patterns. These examinations will be performed 3 times: at the beginning of the trial, after one month and after two months. The trial design is explained in the following paragraph.

The investigators hypothesize that the gait pattern will be improved while using the knee orthosis,as will be expressed by smaller base width and faster walking velocity etc.

DETAILED DESCRIPTION:
The 8-week prospective, randomized controlled study design is depicted in Figure 1. The subjects will be randomly divided into two groups: group A (n=30) or group B (n=30). The patients will be randomly assigned to the study groups , using a block sampling method. The gait pattern, symmetry, and balance of each subject will be evaluated according to the tests described below. After the initial evaluation, group A will be fitted with the Genu Neurexa orthosis for the first four weeks of the study. Group B will not receive treatment for the first four weeks of the study. The subjects will be retested after 4 weeks. Then, group A will ambulate without the Genu Neurexa orthosis for the last 4 weeks. Group B will receive the Genu Neurexa orthosis for the last 4 weeks of the study. Both groups will be retested after 8 weeks for the time of enrollment. This design will provide intra-subject and inter-subject comparison.

The evaluation protocol:

The evaluation tools include subjective patient's satisfactory questionnaire, complete physical and functional evaluation and gait analysis (spatio-temporal parameters and paretic knee angle in the sagittal plane), as well as dynamic electromyography (EMG) muscle activation patterns. The evaluation tools are detailed below.

Gait analysis will be performed while subjects walk on a 6m-long walking path. First, video-recorded observational analysis through the coronal and sagittal planes will be performed in order to register the overall walking pattern and compensation mechanisms.

The main outcome measures will be spatiotemporal parameters (stride time, step time, stance duration, swing duration, double support duration, stride length, step length, base width, toe out angle, cadence and velocity) acquired using 4 markers.

Two-dimensional kinematics examination will be conducted using three markers, located on the paretic limb, in order to measure exact knee angle in the sagittal plane.

The subjects will be instructed to walk several times at their chosen speed on the path, while 4 cameras record the location of the markers. Post analyses, composed of marker identification and tracking (using commercial software by Simi Reality Motion Systems, Germany) and calculations of spatiotemporal parameters, will not be performed in the presence of the subject.

Finally, surface EMG electrodes will be attached to 3 muscles on each leg for dynamic evaluation of dynamic muscle activation pattern during gait. Specifically, we will monitor the gastrocnemius, soleus, and rectus femoris in each leg.

Complete physical evaluation will be conducted to assess range of motion of the joints and muscle tonus.

Functional evaluation of each subject will be accomplished using the Six-Minute Walk Test (6MWT), 10-meter walk test, timed-up-and-go test (TUG) and Berg balance scale (BBS). The BBS is a 14-item scale, designed to measure balance in the clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering a first stro(at least 3 months post stroke)
* Cognitive and cooperative ability to follo instructions.
* Patients suffering from paresis of leg muscles resulting in knee hyperextension.
* Ability to walk with or without a walking aid (cane, walker) independently

Exclusion Criteria:

* Cognitive disorders preventing the subject from understanding the trial protocol, signing a consent form or following the researcher's instructions
* Skin disease or wounds at the paretic knee
* Ankle or foot contructure or limited range of motion
* Orthopaedic injury to the paretic or non-paretic limbs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Spatiotemporal parameters | Up to 3 months
  stride time, step time, stance duration, swing duration, double support duration, stride length, step length, base width, toe out angle, cadence and velocity

SECONDARY OUTCOMES:
Dynamic EMG recordings | Up to 3 months
  Surface EMG electrodes will be attached to 3 muscles on each leg for dynamic evaluation of dynamic muscle activation pattern during gait. Specifically, we will monitor the gastrocnemius, soleus, and rectus femoris in each leg
Sagittal angle of the paretic knee | Up to 3 months
  Sagittal angle of the paretic knee
Functional evaluation | Up to 3 months
  Functional evaluation of each subject will be accomplished using the Six-Minute Walk Test (6MWT), 10-meter walk test, timed-up-and-go test (TUG) and Berg balance scale (BBS). The BBS is a 14-item scale, designed to measure balance in the clinical setting

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel